CLINICAL TRIAL: NCT01270243
Title: Bacterial Microbiota In The Tonsils Of Children Undergoing Adenotonsillectomy And Normal Controls
Brief Title: Bacterial Microbiota In The Tonsils Of Children
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-636-A
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Adenotonsillitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control: No tonsilar or adenoid problems
- Adenotonsillectomy (recurrent): Recurrent adenotonsillitis
- Adenotonsillectomy (obstruction): Upper airway obstruction

SUMMARY:
We, the investigators, propose to look at the bacteria on and in tonsils using gene microarrays. We expect to find previously reported bacteria but also the possibility of previously undetected organisms. We think that the bacterial pathogens present on the tonsillar surface are different from the tonsil core. And we also think that the bacteria of the tonsil surface will differ between patients undergoing adenotonsillectomy and normal controls with no adenotonsillar problems.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for subjects undergoing surgery:

* Age 2-12 yrs
* Both males and females
* Undergoing adenotonsillectomy

Additional criteria for subjects in the recurrent infection group:

* Sleep questionnaire score <5
* Designated by surgeon as having recurrent adenotonsillitis as reason for surgery

Additional criteria for subjects in the airway obstruction group:

* Sleep questionnaire score >5
* Presence of positive polysomnogram desired but not necessary
* Designated by surgeon as having airway obstruction or sleep apnea as reason for surgery

Inclusion criteria for control subjects:

* Age 2-12 yrs
* Both males and females
* No history of adenotonsillar problems
* Sleep questionnaire score < 5

Exclusion Criteria:

Exclusion Criteria for both groups:

* Antibiotic intake in the past 10 days
* Other major medical problems (immune deficiency, cystic fibrosis, malignancy) In the surgery group: designated by surgeon as having both recurrent adenotonsillitis and airway obstruction as reason for surgery Menstruating females

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing adenotonsillectomies at the Comer Children's Hospital
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2017-02-18 (Actual); Study Completion 2017-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fuad M Baroody, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States